CLINICAL TRIAL: NCT04397198
Title: New Imaging-Derived Biomarkers Based On Tridimensional CTA/MRI Hybrid Models For Complex Assessment Of Myocardial Viability After Myocardial Infarction-the HYBRIDHEART Study
Brief Title: The Assessment Of Myocardial Viability Based On CTA/MRI Hybrid Models
Acronym: HYBRIDHEART
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: University of Targu Mures, Romania (Other); Tîrgu Mureș Emergency Clinical County Hospital, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0120-HYBH
Record Dates: First submitted 2020-05-16; First posted 2020-05-21 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2020-05

CONDITIONS: Acute Myocardial Infarction; Myocardial Viability; Vulnerable Coronary Plaques; Coronary Stenosis; Myocardial Fibrosis
Keywords: biomarkers; myocardial infarction; hybrid images; myocardial viability; CCTA; MRI
MeSH Terms: conditions — Coronary Stenosis; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood samples for evaluation of the level of hs-CRP, myocardial necrosis markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIBRIDH-SG 01: Study subjects with documented ST segment Elevation Myocardial Infarction
  Interventions: Diagnostic Test: Speckle Tracking echocardiography

INTERVENTIONS:
Diagnostic Test: Speckle Tracking echocardiography — Diagnostic tests:
  Speckle Tracking echocardiography with analyzing the myocardial strain, myocardial velocities, 128-multislice CCTA with the evaluation of the Calcium Scoring (total and local) , identifying the coronary stenosis, evaluation of the plaque vulnerability degree, assess polar maps of the myocardium.
  MRI for the evaluation of the percentage of myocardial scar, also the percentage of the viable myocardial tissue using contrast late enhancement sequences, measuring myocardial fibrosis using Q-mass software.
  Diagnostic tests:
  Laboratory assessment for the evaluation of the level of hs-CRP and myocardial necrosis biomarkers
  Other Names: 128-multislice CCTA; MRI; Laboratory assessment

SUMMARY:
The aim of HYBRIDHEART study is to develop new imagistic prototype for a complex evaluation of the myocardial viability by superposing computed tomographic angiographic polar maps of the myocardium with magnetic resonance imaging contractile maps in subjects who suffered an acute myocardial infarction. Moreover, the study will evaluate the association of myocardial viability with the level of inflammatory markers and the percent of myocardial fibrosis, also will correlate the imaging-derived parameters with the inflammatory status of the patients, left ventricular function, ischemic time and major adverse cardiovascular events (MACE) rate.

DETAILED DESCRIPTION:
The HYBRIDHEART study is a prospective, observational study that will be conducted in the Laboratory of Advanced Research in Cardiac Multimodal Imaging of Cardio Med Medical Center Tîrgu Mureş, Romania.

The project will include 100 subjects with documented ST Segment elevation myocardial infarction at 30 days prior to study enrollment. The level of inflammatory biomarkers will be express using hs-CRP levels at day 1 and day 5 post the acute event. All the subjects will undergo coronary computer tomography angiography (CCTA), magnetic resonance (MRI), 3D contrast enhancement echocardiography, speckle tracking echocardiography at the moment of the inclusion. Also, venous blood samples will be collected for the determination of the level of hs-CRP and myocardial necrosis biomarkers such as I Troponin, myocardial fraction of creatine kinase (CK-MB).

The imagistic acquisitions obtained from all the techniques used, will be processed using a supercomputer set up with computational simulations applications for the myocardial kinetics. All the MRI images will be analyzed using Medis Q-mass software in order to quantify the myocardial fibrosis, and the CCTA images will be analyzed using SyngoVia. Frontier software, for the plaques evaluation. The images will be superposed obtaining hybrid CCTA-MRI images that will be analyzed in order to correlate the degree of plaque vulnerability, the percent of myocardial scar, the percent of viable myocardial tissue, calculating the total Calcium Scoring, Syntax score.

The study will be conducted over a period of 2 years, in which the subjects will be examined at the moment of inclusion and during the follow-up visits. Will be performed the follow up of the subjects at 1, 3 and 6 months and 1 year after the inclusion period. At 1 month follow up the subjects will be examined, will be performed echocardiography. Moreover during follow up will be done telephonic visits with target questions . MACE rate will be assessed at 6 month follow-up and 1 year follow up visits.

Study objectives:

Primary: to develop new imagistic markers for a complex evaluation of the myocardial viability, by superposing computed tomographic angiographic polar maps of the myocardium with MRI contrast enhancement maps in subjects with myocardial infarction.

Secondary: to evaluate the association of the percent of viable myocardium with the level of inflammatory markers. To correlate the plaque vulnerability markers with the percent of myocardial fibrosis, the inflammatory status of the subjects, left ventricular function, ischemic time and the rate of MACE, Calcium Score, Syntax score

Study timeline:

Baseline (day0) Obtain a written consent from the participants on study consent form. Verify inclusion/exclusion criteria Assess the demographical data of the participants, medical history, possible known allergies, medication history, alcohol, tobacco use history Physical examination record Blood pressure record 12-lead ECG Collect venous blood samples Performing CCTA, MRI, Speckle Tracking Echocardiography using standard protocols

Visit 1 (month 1) Physical examination record 12-lead ECG Blood pressure record Transthoracic Echocardiography

Visit 2 (month 3) Telephone visit with target questions, all the answers recorded in study forms.

Visit 3 (month 6) End point evaluation 12-lead ECG Blood pressure record Transthoracic Echocardiography

Visit 4 (12 months) End point evaluation 12-lead ECG Blood pressure record Transthoracic Echocardiography Performing CCTA

Study procedures:

Clinical examinations 12 lead ECG Laboratory assessment for the evaluation of the level of hs-CRP and myocardial necrosis biomarkers (I Troponin, CK-MB) Speckle Tracking echocardiography with analyzing the myocardial strain, myocardial velocities, left ventricular function 128-multislice CCTA with the evaluation of the Calcium Scoring (total and local) , identifying the coronary stenosis, evaluation of the plaque vulnerability degree, assess polar maps of the myocardium.

MRI for the evaluation of the percentage of myocardial scar, also the percentage of the viable myocardial tissue using contrast late enhancement sequences, measuring myocardial fibrosis using Q-mass software.

Data collection:

A dedicated database will be created, including all the demographical data and data regarding the acute myocardial infarction, such as: infarct location, time of ischemia, ECG changes, levels of the necrosis markers, hs-CPR, MRI findings, CCTA findings, speckle tracking parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old
* Patients with documented ST segment Elevation Myocardial Infarction in the last 30 days
* Patients who signed the written consent.

Exclusion Criteria:

* Subjects with renal impairment, or contrast intolerance
* Pregnant women
* Patients known with malignancy in the last year
* Non-compliant patients
* Patients older than 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 subjects with documented ST Segment elevation myocardial infarction at 30 days prior to study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Hybrid imaging | 6 months
  the development of the new hybrid imaging features: plaque vulnerability degree, % of myocardial scar, % of viable myocardial tissue

SECONDARY OUTCOMES:
Correlations | 12 months
  Association of the level of hs-CRP in relation with MACE rate, time of ischemia, myocardial viability, percent of myocardial fibrotic tissue, plaque vulnerability degree and left ventricular function

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio Med, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD sharing time is starting 6 months after the publication.